CLINICAL TRIAL: NCT06364462
Title: Establishment of Precise Evaluation Criteria for Histological Regression of NASH-related Liver Fibrosis
Brief Title: Precise Evaluation Criteria for Histological Regression of NASH Fibrosis
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jidong Jia, Principal Investigator, Beijing Friendship Hospital
Other Study IDs: ZLRK202301
Record Dates: First submitted 2024-03-12; First posted 2024-04-15 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: NASH; Liver Fibrosis
Keywords: NASH; Liver fibrosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group of NASH-related liver fibrosis
  Interventions: Other: lifestyle intervention

INTERVENTIONS:
Other: lifestyle intervention — Dietary recommendations should consider energy restriction and exclusion of MAFLD-mediating components (processed food, food and beverages high in added fructose). A Mediterranean type diet is advisable. Both aerobic exercise and resistance training effectively reduce liver fat and should be tailored based on patient preferences to ensure long-term adherence.

SUMMARY:
It is an observational study of NASH patients with a calculated sample size of 220. Liver biopsy-proven NASH fibrosis with stage F2-F4 will be recruited in this study. A second biopsy will be performed after clinical trials or 1-3 years of lifestyle intervention. Patients will be followed up at baseline and every six months with h-CRP, liver function tests, fasting blood glucose, fasting insulin, ferritin, liver ultrasonography, and liver stiffness measurements.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age.
* Liver biopsy-proven NASH fibrosis with stage F2-4.
* Signature of written informed consent.

Exclusion Criteria:

* Patients with other liver diseases, including viral hepatitis, alcoholic liver diseases, autoimmune liver diseases, genetic metabolic liver disease, drug-induced liver diseases, and infected with HIV.
* Pregnant women.
* Patients have the following conditions before liver biopsy:

Hepatocellular carcinoma or suspected liver cancer; Decompensated cirrhosis: including ascites, hepatic encephalopathy, esophageal variceal bleeding, hepatorenal syndrome; Other malignancy; Undergone liver transplantation surgery;

* Patients with any other reasons not suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NASH patients with fibrosis stage F2-4 diagnosed with liver biopsy
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2027-03-09 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Regression of NASH fibrosis | 1-3 years
  Regression of NASH fibrosis based on liver biopsy

SECONDARY OUTCOMES:
Dynamic changes of liver stiffness measurements (LSM) | 3 years
  Dynamic changes of liver stiffness measurements (LSM)
Dynamic changes of Controlled Attenuation Parameter (CAP) | 3 years
  Dynamic changes of CAP, higher scores mean a worse outcome.
Dynamic changes of Magnetic Resonance Elastography (MRE) | 3 years
  Dynamic changes of MRE, higher scores mean a worse outcome.
Dynamic changes of Magnetic Resonance Imaging Proton Density Fat Fraction (MRI-PDFF) | 3 years
  Dynamic changes of MRI-PDFF, higher scores mean a worse outcome.
Dynamic changes of non-invasive liver fibrosis models | 3 years
  Dynamic changes of Aspartate Aminotransferase to Platelet Ratio Index (APRI), , higher scores mean a worse outcome.
Dynamic changes of non-invasive liver fibrosis models | 3 years
  Dynamic changes of Fibrosis-4 Index (FIB-4), higher scores mean a worse outcome.
Dynamic changes of non-invasive liver fibrosis models | 3 years
  Dynamic changes of BARD (BMI, AST/ALT Ratio, Diabetes), higher scores mean a worse outcome.
Dynamic changes of non-invasive liver fibrosis models | 3 years
  Dynamic changes of NAFLD Fibrosis Score (NFS), higher scores mean a worse outcome.
Dynamic changes of non-invasive liver fibrosis models | 3 years
  Dynamic changes of FibroScan-aspartate aminotransferase score (FAST), higher scores mean a worse outcome.
Dynamic changes of metabolic markers | 3 years
  Dynamic changes of Body Mass Index (BMI), higher scores mean a worse outcome.
Dynamic changes of metabolic markers | 3 years
  Dynamic changes of fasting glucose
Dynamic changes of metabolic markers | 3 years
  Dynamic changes of serum lipid level
Incidence of liver-related events | 3 years
  Incidence of ascites, hepatic encephalopathy, esophageal variceal bleeding, hepatocellular carcinoma, liver-related death/liver transplantation
Incidence of extrahepatic related events | 3 years
  Incidence of cardiovascular and cerebrovascular events, extrahepatic malignancies, metabolic diseases

CONTACTS AND LOCATIONS:
Overall Officials: Jidong Jia, Professor, Principal Investigator — Beijing Friendship Hospital; Jingmin Zhao, Professor, Principal Investigator — Beijing 302 Hospital; Jing Zhang, Principal Investigator — Beijing You-an Hospital, Capital Medical University; Minghui Li, Principal Investigator — Beijing Ditan Hospital

IPD SHARING:
Plan to Share IPD: Undecided